CLINICAL TRIAL: NCT00804505
Title: A 90 Day Multi-Center, Randomized, Parallel Group Daily Wear Investigation of a New Hybrid Lens SynergEyes SA Manufactured With a Rigid Gas Permeable Center (Petrafocon A) and a Silicone Hydrogel Skirt (Larafilcon A) Compared to SynergEyes A (Paflufocon D Hem-iberfilcon A)
Brief Title: Hybrid SA RGP Center/S-H Skirt Daily Wear 90 Day Multicenter Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SynergEyes, Inc. (Industry)
Responsible Party: SynergEyes, Inc., Joe Collins
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SI-0804 V1.0
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Corneal Disease; Hypersensitivity
Keywords: Substantial equivalence to control device
MeSH Terms: conditions — Corneal Diseases; Hypersensitivity | interventions — Contact Lenses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Test arm daily wear hybrid contact lens.
  Interventions: Device: SynergEyes Hybrid (petrafocon A hem-larafilcon A) Hybrid Contact Lens
- 2 (Other): Control: SynergEyes Hybrid (paflufocon D hem-iberfilcon A) Hybrid Contact Lens
  Interventions: Device: SynergEyes Hybrid (paflufocon D hem-iberfilcon A) Contact Lens

INTERVENTIONS:
Device: SynergEyes Hybrid (petrafocon A hem-larafilcon A) Hybrid Contact Lens — Comparison to control hybrid lens with similar 'dose'minimum 8 hours daily use for up to 90 days.
  Arms: 1
Device: SynergEyes Hybrid (paflufocon D hem-iberfilcon A) Contact Lens — Comparison to test lens: Daily use for minimum 8 hours up to 90 days.
  Arms: 2

SUMMARY:
The purpose of the study is to demonstrate that the SynergEyes SA Hybrid Contact Lens clinical performance is substantially equivalent to that of the SynergEyes A Hybrid Lens when studied:

* within the corresponding range of lens powers
* in a population randomized within multiple investigational sites
* with a study ration of 2/1 test vs control lenses
* for a duration of 90 days.

DETAILED DESCRIPTION:
The objective of the study is to compare the SynergEyes SA Hybrid Contact Lens (Test) to the SynergEyes A Hybrid Contact lens (Control) when used in a daily wear regimen on non-diseased eyes for the correction of myopia (-0.25 to -6.00Diopters) with up to -2.50 Diopters of astigmatism. The population will be randomized into a 2/1 ratio of the Test/Control for 90 days. The study objective is to complete at least 40 subjects in the Test material and 20 subjects in the Control material.

The purpose of the study is to demonstrate that the SynergEyes SA Hybrid Contact Lens clinical performance is substantially equivalent to that of the SynergEyes A Hybrid Lens when studied within the corresponding range of powers in a population randomized within investigational sites to produce a 2/1 ratio of Test vs. Control lenses.

ELIGIBILITY:
Inclusion Criteria:

Prior to being considered eligible to participate in this study, each subject MUST:

1. Be at least 18 years of age as of the date of evaluation.
2. Have

   1. read the Informed Consent,
   2. been given an explanation of the Informed Consent,
   3. indicated an understanding of the Informed Consent and
   4. signed the Informed Consent Form.
3. Be willing and able to adhere to the instructions set forth in this protocol and able to keep all specified appointments.
4. Be a current contact lens wearer.
5. Possess wearable and visually functional eyeglasses.
6. Be in good general health, based on his/her knowledge.
7. Require spectacle lens powers between plano and -6.00 diopters sphere with no more than -2.50 diopters of spectacle refractive astigmatism and be willing to wear lenses in both eyes.
8. Have manifest refraction visual acuity equal to or better than 20/25 in each eye.

Exclusion Criteria:

* Subjects may not be enrolled into the study if ANY of the following apply:

  1. Subject is wearing lenses in a monovision modality and is unwilling to be fit with distance lenses in both eyes. NOTE: Subjects may NOT wear monovision lenses at any time during the study as it will interfere with the distance visual acuity measurement.
  2. Subject exhibits poor personal hygiene.
  3. Subject is currently or within 30 days prior to this study has been an active participant in another clinical study.
  4. Subject is currently pregnant (to the best of the subject's knowledge), is planning a pregnancy within the next 3 months or is lactating.
  5. Subject is a member, relative or household member of the office staff, including the investigator(s).
  6. Subject has a known sensitivity to ingredients used in contact lens care products or over-the-counter lubricants and artificial tears.
  7. Subject has undergone refractive surgery or is currently receiving or has previously received orthokeratology treatment.
  8. Subject is aphakic or pseudophakic.
  9. Subject has ocular or systemic disease such as, but not limited to: anterior uveitis or iritis (past or present), glaucoma, Sjögren's syndrome lupus erythematosus, scleroderma, keratoconus or type II diabetes.
  10. Use of ocular medications for any reason or systemic medications which might interfere with contact lens wear.
  11. A known history of corneal hypoesthesia (reduced corneal sensitivity).
  12. Slit lamp findings that would contraindicate contact lens wear, including but not limited to:

      * History of corneal ulcer, corneal infiltrates or fungal infections
      * Corneal scars within the visual axis
      * Pterygium
      * Dry eye symptoms with decrease tear levels and punctate staining ≥ Grade 2
      * Neovascularization or ghost vessels > 1.5 mm in from the limbus
      * Seborrhoeic eczema, seborrhoeic conjunctivitis
      * History of papillary conjunctivitis that has interfered with lens wear or a current condition of Grade 2 (Mild) or greater
  13. Clinically significant (Grade 3 or 4) anterior segment abnormalities or any infection of the eye, lids, or associated structures.

TO BE ELIGIBLE TO BE RANDOMIZED FOR STUDY PRODUCT TRIAL A SUBJECT MUST HAVE ALL OF THE INCLUSION CRITERIA AND NONE OF THE EXCLUSION CRITERIA PRESENT.

TO BE ELIGIBLE FOR LENS DISPENSING, THE SUBJECT'S STUDY DEVICE CONTACT LENS VISUAL ACUITY MUST BE EQUAL TO OR BETTER THAN 20/30 IN EACH EYE

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2008-06; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Comparison of objective findings (slit lamp, lens fitting, deposits, subjective symptoms, adverse events test vs control | 3 months
Visual acuity comparison test/control. | 3 mo.

CONTACTS AND LOCATIONS:
Overall Officials: William Gleason, OD, Study Director — Foresight Regulatory Strategies, Inc.
Locations (8):
- United States (8):
  - Carmel Mountain Vision Care, San Diego, California
  - Silicon Valley Eye Physicians, Sunnyvale, California
  - Casazza Optometric Group, Andover, Massachusetts
  - Vision Care Associates, East Lansing, Michigan
  - Western Reserve Vision Care, Inc., Beachwood, Ohio
  - Dr. Karambelas & Associates, Providence, Rhode Island
  - Primary Eyecare Group P.C., Brentwood, Tennessee
  - Snowy Range Vision Center, Laramie, Wyoming